CLINICAL TRIAL: NCT05708768
Title: Developing and Implementing Digital, Innovative, Sustainable, and Knowledge-based Municipal Healthcare Services in Acute Illness and Trauma
Brief Title: Digital, Innovative, Sustainable, and Knowledge-based Acute Municipal Healthcare Services Illness and Trauma
Status: Completed | Type: Observational
Sponsor: Ostfold University College (Other)
Collaborators: Oslo University Hospital (Other); Ostfold Hospital Trust (Other); OsloMet (Unknown)
Responsible Party: Sponsor
Other Study IDs: 971 567 376
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Multiple Chronic Conditions; Acute Disease
MeSH Terms: conditions — Multiple Chronic Conditions; Acute Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Acutely ill persons in the municipality: Patients recieving services from a rapid response vehicle manned with dedicated physicians from the municipality
  Interventions: Other: Receiving physician manned rapid response car services

INTERVENTIONS:
Other: Receiving physician manned rapid response car services — All patients receiving services from the physician manned rapid response car will be included

SUMMARY:
Through introducing physicians in front in the medical assessment and decision-making processes in acute and sub-acute illness in the municipalities, as well as including machine learning in analyzing prospective and retrospective data, the project will develop and implement innovative and knowledge-based digital diagnostic tools and decision-making support systems to be used in the municipalities. As such, the project will contribute to early identification of severe illness, prevent deterioration of disease, and facilitate early medical intervention.

DETAILED DESCRIPTION:
The overall objective of the project is to determine if and how innovative digital decision-making tools based on artificial intelligence (AI) can help to develop more accessible, efficient, cost-effective, and sustainable municipal healthcare services. More specifically, the project aims are:

* to explore different outcomes of a municipal rapid response car manned with dedicated physicians
* to compare outcomes from Norwegian and Swedish out-of-hospital EMS in acute illness
* to explore how decision-making tools based on AI can be used to optimize dispatch
* to explore how decision-making tools based on AI can assist dispatched personnel and in prehospital care
* to determine the quality and efficacy of the different systems explored through cost-analyses and exploration of stakeholders' experiences with the decision-making tools

ELIGIBILITY:
Inclusion Criteria:all patients receiving services from the physician manned rapid response car -

Exclusion Criteria:none

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients recieving services from the physician manned rapid response car will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
At location | 2 hours
  Patients treated at location

SECONDARY OUTCOMES:
Transported | 2 hours
  Patients being transported for further diagnostics

OTHER OUTCOMES:
Institutionalized | 12 hours
  Patients being institutionalized

CONTACTS AND LOCATIONS:
Overall Officials: Randi M Sommerfelt, PhD, Study Chair — Østfold University College
Locations (1):
- Fredrikstad Casualty, Fredrikstad, Akershus, Norway

IPD SHARING:
Plan to Share IPD: Yes
The goal is to publish anonymized datasets. ØUC is an institutional member of the DataverseNO community in Norway, and the DataverseNO-based repository ØUC Open Research Data, which is a generic repository of high quality, is suitable for this endeavor. A part of the data generated by this research project consists of qualitative interviews. In case these data cannot be anonymized, open publication of data will be refrained and rather opt for making metadata available. Datasets and metadata will be published in connection with open access publication of research articles.
Supporting Information: Study Protocol, CSR
Time Frame: After all publication